CLINICAL TRIAL: NCT03153085
Title: A Phase II Study of Combination Treatment with TBI-1401(HF10), a Replication-competent HSV-1 Oncolytic Virus, and Ipilimumab in Japanese Patients with Stage IIIB, IIIC, or IV Unresectable or Metastatic Malignant Melanoma
Brief Title: A Study of Combination with TBI-1401(HF10) and Ipilimumab in Japanese Patients with Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI1401-02
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
Keywords: Unresectable melanoma; Metastatic melanoma; Recurrent Melanoma; TBI-1401(HF10); HF10; HSV-1; Oncolytic virus; Oncolytic viral immunotherapy; Ipilimumab; Intratumoral administration; canerpaturev
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBI-1401(HF10) + Ipilimumab (Experimental): 1x10^7 TCID50/mL TBI-1401(HF10) administered to a single or multiple eligible tumors in a total volume up to 5.0 mL (injection volume will be adjusted based on the size of tumor mass) by intratumoral injection and 3 mg/kg ipilimumab administered by intravenous infusions.
  Interventions: Biological: TBI-1401(HF10); Drug: Ipilimumab

INTERVENTIONS:
Biological: TBI-1401(HF10) — 1x10^7 TCID50/mL TBI-1401(HF10) (for a total of 6 injections; the first 4 injections at 1-week intervals; the remaining 2 injections at 3-week intervals).
  Following combination therapy, patients may continue to receive the 1x10^7 TCID50/mL TBI-1401(HF10) alone for up to an additional 13 injections (total of 19 injections = 1 year) if eligible for administration.
  Other Names: HF10; canerpaturev
Drug: Ipilimumab — 3 mg/kg ipilimumab (for a total of 4 intravenous infusions, each administered at 3-week intervals).
  Other Names: anti CTLA-4 antibody

SUMMARY:
The purpose of this study is to determine if TBI-1401(HF10) in combination with ipilimumab is effective in Japanese patients with stages IIIB, IIIC, or IV unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
The study is designed to assess efficacy and safety with repeated administration of intratumoral injections of TBI-1401(HF10) at 1x10^7 TCID50/mL in combination with intravenous infusions of 3mg/kg ipilimumab in Japanese patients.

This is a single arm, open label Phase II study, to evaluate the efficacy and safety of TBI-1401(HF10) treatment in combination with the immunologic checkpoint inhibitor, ipilimumab (anti-CTLA-4 monoclonal antibody). The study population will include patients with Stage IIIB, IIIC or IV unresectable or metastatic malignant melanoma who are ipilimumab-eligible.

Patients will receive the dose of 1x10^7 TCID50/mL TBI-1401(HF10) (for a total of 6 injections; the first 4 injections at 1-week intervals; the remaining 2 injections at 3-week intervals) + ipilimumab at 3 mg/kg (for a total of 4 intravenous infusions, each administered at 3-week intervals).

Following combination therapy, patients may continue to receive the 1x10^7 TCID50/mL TBI-1401(HF10) alone for up to an additional 13 injections (total of 19 injections = 1 year) if they have tolerated the study treatment, are responding, have stable disease, or have progressive disease that is not clinically significant in the judgment of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed Stage IIIB, IIIC or IV unresectable or metastatic melanoma except uveal melanoma, who must have a history of treatment (chemotherapy, molecular targeted therapy, or anti PD-1 antibody therapy).
* Patients must have measurable non-visceral lesion(s) that are evaluable by the modified World Health Organization (mWHO) criteria and immune-related response criteria (irRC).
* Patients must be ≥ 20 years of age.
* Patients must have a life expectancy ≥ 24 weeks.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Patients must have adequate organ function, defined as

  * Total bilirubin levels ≤ 1.5 x upper limit of normal [ULN] (except for patients with Gilbert's Syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
  * AST/ALT levels ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present.
  * Creatinine ≤ 1.5 x ULN or creatinine clearance (calculated) ≥ 60 mL/min/1.73 m^2 for patients with creatinine > 1.5 x ULN.
  * Absolute neutrophil count ≥1,500/µL and
  * Platelet count ≥ 75,000/ µL
* Men and women of childbearing potential must agree to use adequate contraception from the time of consent through 30 days after final study treatment.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 1 week prior to start of treatment.
* Patients must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients who were previously treated with ipilimumab by intravenous infusion.
* Patients receiving chemotherapy or molecularly targeted drug or anti-PD-1 antibody treatment or radiotherapy or immunotherapy within 4 weeks prior to initiating study treatment.
* Patients with a history of Grade 4 adverse events caused by chemotherapy, molecularly targeted drug, anti-PD-1 antibody treatment, radiotherapy or immunotherapy conducted more than 4 weeks prior to TBI-1401(HF10) treatment, or presence of such adverse events of Grade 2 or greater, except alopecia and adverse events controlled by a treatment.
* Patients receiving anti-herpes medication within 1 week prior to initiating TBI-1401(HF10) administration, except local treatment such as ointment.
* Patients with a history of significant tumor bleeding, or coagulation or bleeding disorders.
* Patients with target tumors that could potentially invade a major vascular structure (e.g., innominate artery, carotid artery), based on unequivocal imaging findings.
* Patients with Grade 2 or greater neurologic abnormalities (CTCAE version 4.0), including Grade 2 or greater peripheral neuropathy caused by previous treatments.
* Patients with clinically evident Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C virus (HCV), or Epstein-Barr virus (EBV) infection.
* Patients requiring systemic glucocorticoid (except 10 mg/day/body prednisolone or less) or immunosuppressive therapy because of the presence or history of autoimmune disease (e.g., Crohn's disease, ulcerative colitis) or other diseases.
* Concurrent use of any other investigational agents within 4 weeks prior to initiating study treatment.
* Patients with active CNS metastases or carcinomatous meningitis, except patients with CNS lesions that have been treated and have no evidence of progression in the brain on CT/MRI for ≥ 3 months.
* Pregnant or breastfeeding women (excluding the case in which breastfeeding is discontinued and will not resume it); women desiring to become pregnant within the timeframe of the study are also excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Best overall response rate (BORR) by irRC | at 24 weeks
  Determine the efficacy of TBI-1401(HF10) in combination with Ipilimumab evaluated by irRC (immuno-related response criteria)

SECONDARY OUTCOMES:
Best overall response rate (BORR) by mWHO response criteria | at weeks 24
  Determine the efficacy of TBI-1401(HF10) in combination with Ipilimumab evaluated by modified WHO (mWHO) response criteria
Best overall response rate (BORR) by RECIST version 1.1 | at weeks 24
  Determine the efficacy of TBI-1401(HF10) in combination with Ipilimumab evaluated by RECIST version 1.1
Objective response rate (ORR) by irRC | at weeks 6, 12, 18, and 24
  Overall tumor response evaluated by irRC in the measurable target lesion(s) and unmeasurable/evaluable target lesion(s).
Objective response rate (ORR) by mWHO | at weeks 6, 12, 18, and 24
  Overall tumor response evaluated by mWHO response criteria in the measurable target lesion(s) and unmeasurable/evaluable target lesion(s).
Objective response rate (ORR) by RECIST version 1.1 | at weeks 6, 12, 18, and 24
  Overall tumor response evaluated by RECIST version 1.1 in the measurable target lesion(s) and unmeasurable/evaluable target lesion(s).
Adverse event summaries, vital signs, and laboratory parameters to evaluate the safety and tolerability. | through study completion, up to 1 year
  Adverse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.0).
Progression-free survival (PFS) | through disease progression, up to 3 years
  Evaluation the time to progression during and after the treatment.
Durable response rate (DRR) | for 1 year
  Evaluation the length of time after a partial or complete response.
1 year survival rate | at 1 year
  Determine the 1 year survival rate of patient who received treatment.

OTHER OUTCOMES:
Levels of antibody to HSV-1 | up to weeks 24
  Evaluate the change of anti-HSV-1 antibody levels.
Change in immunologic parameters in serum | up to weeks 24
  Analysis the change of cytokine profiles, antitumor T-cell reactivity and regulatory T-cell (Treg) population by immunoassay and flow cytometry.
Histopathological response with TBI-1401(HF10) administrated tumor | up to weeks 24
  Biopsies will be performed to evaluate the histopathological response with TBI-1401(HF10) administrated tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Naoya Yamazaki, Principal Investigator — National Cancer Center Hospital
Locations (12):
- Japan (12):
  - Clinical Site, Nagakute, Aichi-ken
  - Clinical Site, Nagoya, Aichi-ken
  - Clinical Site, Fukuoka, Fukuoka
  - Clinical Site, Kurume, Fukuoka
  - Clinical Site, Sapporo, Hokkaido
  - Clinical Site, Tsukuba, Ibaraki
  - Clinical Site, Kumamoto, Kumamoto
  - Clinical Site, Niigata, Niigata
  - Clinical Site, Osaka, Osaka
  - Clinical Site, Shizuoka, Shizuoka
  - Clinical Site, Chūōku, Tokyo
  - Clinical Site, Chūō, Yamanashi

IPD SHARING:
Plan to Share IPD: No